CLINICAL TRIAL: NCT01070043
Title: A Single Center, Randomized, Double-blind, Active Controlled, Parallel Group Study to Demonstrate Non-inferiority of a Fixed Dose Combination of 5 mg Amlodipine and 80 mg Valsartan to 160 mg Valsartan in the Treatment of Hypertension
Brief Title: To Demonstrate Non-inferiority of Combination of 5 mg Amlodipine/ 80 mg Valsartan to 160 mg Valsartan Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAA489ATW01
Record Dates: First submitted 2010-02-06; First posted 2010-02-17 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension; High Blood Pressure
Keywords: Hypertension; valsartan; amlodipine; high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Valsartan; Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amlodipine 5mg/Valsartan 80 mg (Experimental): During double-blind treatment period, patients randomized to combination therapy received daily one dosage (Amlodipine/Valsartan 5mg/80mg) with one single tablet size for 8 weeks.
  Interventions: Drug: Amlodipine 5mg/Valsartan 80 mg
- Valsartan 160 mg (Active Comparator): In double blinded treatment period, patients randomized to this arm received 160 mg Valsartan once daily for 8 weeks.
  Interventions: Drug: Valsartan
- Run-In Valsartan 80 mg (Other): During run-in period, oral valsartan 80 mg once daily for 4 weeks.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Amlodipine 5mg/Valsartan 80 mg — Combination therapy of Amlodipine/Valsartan 5mg/80mg one dosage daily with one single tablet size for 8 weeks.
  Other Names: Exforge
  Arms: Amlodipine 5mg/Valsartan 80 mg
Drug: Valsartan — For run-in period, Valsartan 80 mg daily in one dosage with one single tablet size for 4 weeks.
  Monotherapy for double blind treatment period in one dosage (Valsartan 160mg) daily with one single tablet size for 8 weeks
  Other Names: Diovan
  Arms: Run-In Valsartan 80 mg; Valsartan 160 mg

SUMMARY:
The purpose of the study was to assess efficacy and safety of fixed dose combination of 5 mg amlodipine/80 mg valsartan compared to 160 mg valsartan monotherapy in lowering blood pressure in Taiwanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years of age with hypertension defined as sitting systolic blood pressure between 140 mmHg and 180 mmHg or sitting diastolic blood pressure between 90 mmHg and 120 mmHg.
* High risk participants ( defined as having: (diabetes mellitus, chronic renal disease, Framingham 10-year risk score >10%, established coronary artery disease (CAD), or CAD equivalents including carotid artery disease, peripheral arterial disease (PAD), abdominal aortic aneurysm (AAA))with hypertension defined as sitting systolic blood pressure between 130 mmHg and 180 mmHg or sitting diastolic blood pressure between 80 mmHg and 120 mmHg.

Exclusion Criteria:

* Known or suspected secondary hypertension
* Known New York Heart Association (NYHA) functional class IV Heart Failure
* History of myocardial infarction, transient ischemic attack or cerebrovascular accident within the preceding 3 months
* Clinically significant valvular disease
* Women who are pregnant, intend to become pregnant or are breastfeeding
* Participants who have severe medical condition(s) that in the view of the Investigator prohibits participation in the study
* Participants who have hypersensitivity to the investigational/ reference drug or any of the components in the formulation.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Novartis, Study Chair — Novartis
Locations (1):
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 4 week run-in phase preceded the randomized, double-blind treatment phase of the study. During the run-in phase, participants took valsartan 80 mg daily before a meal. Sixty participants entered the run-in phase. Those participants who met the inclusion criteria entered the randomized, double-blind treatment phase.
Groups:
- Amlodipine 5 mg/Valsartan 80 mg: During double-blind treatment period, patients randomized to combination therapy received daily one dosage (Amlodipine/Valsartan 5mg/80mg) with one single tablet size for 8 weeks.
Period: Run-In Phase
Arm/Group | Run-In Valsartan 80 mg | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Started | 60 | 0 (This combination therapy arm is used only for double-blind phase.) | 0 (This monotherapy (Valsartan 160 mg) treatment arm is used only for double-blind phase.)
Completed | 42 | 0 | 0
Not Completed | 18 | 0 | 0
Not completed — Did not Meet Inclusion Criteria | 18 | 0 | 0
Period: Double-Blind Treatment
Arm/Group | Run-In Valsartan 80 mg | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Started | 0 | 21 | 21
Completed | 0 | 21 | 19
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine 5mg/Valsartan 80 mg | Valsartan 160 mg | Total
Number analyzed (Participants) | 21 | 21 | 42
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measurements were based on safety/intent-to-treat (ITT) population.
  years | 59.50 (13.81) | 55.13 (11.81) | 57.31 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) From Office Blood Pressure Measurement
Description: Two arterial blood pressure (BP) determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in mean sitting systolic blood pressure (msSBP) was calculated comparing the Week 8 readings to the readings taken at baseline.
Time Frame: Baseline and 8 weeks
Population: The Intent-to-Treat (ITT) Population includes all participants having taken at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 21 | 21
mmHg
  Baseline | 150.26 (12.91) | 141.14 (12.71)
  8 weeks | 133.79 (14.63) | 133.68 (12.73)
  Change from baseline to 8 weeks | -16.48 (15.53) | -7.23 (11.60)

2. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) From Office Blood Pressure Measurement
Description: Two arterial blood pressure (BP) determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in mean sitting diastolic blood pressure (msDBP) was calculated comparing the Week 8 readings to the readings taken at Baseline.
Time Frame: Baseline and 8 weeks
Population: The Intent-to-Treat (ITT) Population includes all participants having taken at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 21 | 21
mmHg
  Baseline | 92.12 (10.84) | 89.98 (9.37)
  8 weeks | 82.29 (8.74) | 86.73 (9.10)
  Change from baseline to 8 weeks | -9.83 (7.66) | -2.65 (6.75)

3. Secondary Outcome: Change From Baseline in Mean Systolic Blood Pressure (mSBP) From Ambulatory Blood Pressure Measurement (ABPM) Over 24 Hours
Description: Validated automated ambulatory blood pressure monitors were dispensed to participants with instructions on correct use. Automated blood pressure readings were obtained every 15-30 minutes during waking hours and every 30-60 minutes during sleep for a total of 24 hours. The change in mean systolic blood pressure (mSBP) over 24 hours was measured from baseline to 8 weeks of treatment during the double-blind phase.
Time Frame: Baseline and 8 weeks
Population: The Intent-to-Treat (ITT) Population includes all participants having taken at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 21 | 21
mmHg
  Baseline | 144.38 (17.39) | 139.76 (13.46)
  8 weeks | 129.67 (14.03) | 131.11 (12.39)
  Change from baseline to 8 weeks | -14.71 (11.64) | -6.39 (12.06)

4. Secondary Outcome: Change From Baseline in Mean Diastolic Blood Pressure (mDBP) From Ambulatory Blood Pressure Measurement (ABPM) Over 24 Hours After 8 Weeks of Treatment During the Double-blind Phase
Description: Validated automated ambulatory blood pressure monitors were dispensed to participants with instructions on correct use. Automated blood pressure readings were obtained every 15-30 minutes during waking hours and every 30-60 minutes during sleep for a total of 24 hours. The change in mean diastolic blood pressure (mDBP) over 24 hours was measured from baseline to 8 weeks of treatment during the double-blind.
Time Frame: Baseline and 8 weeks
Population: The Intent-to-Treat (ITT) Population includes all participants having taken at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 21 | 21
mmHg
  Baseline | 86.95 (14.14) | 87.90 (9.44)
  8 weeks | 79.29 (10.70) | 82.94 (8.42)
  Change from baseline to 8 weeks | -7.67 (7.43) | -3.56 (7.70)

5. Secondary Outcome: Number of Participants With Adverse Events During Double-blind Phase
Time Frame: 8 weeks
Population: Safety population included all patients who received at least one study medication during the study period.
Measure: Number; unit: Participants
Arm/Group | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Number analyzed (Participants) | 21 | 21
Participants
  Total AE | 9 | 15
  At least one AE | 7 | 11
  AE Not related to drug | 9 | 15

ADVERSE EVENTS:
Description: All patients who received at least one study medication during the double-blinded study period were included in the reported safety population.
Arm/Group | Amlodipine 5 mg/Valsartan 80 mg | Valsartan 160 mg
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/21
Other Adverse Events (participants affected / at risk) | 6/21 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5 mg/Valsartan 80 mg (N=21) | Valsartan 160 mg (N=21)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5 mg/Valsartan 80 mg (N=21) | Valsartan 160 mg (N=21)
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.